CLINICAL TRIAL: NCT01177982
Title: Reinforcement-Based Treatment for Pregnant Drug Abusers
Acronym: HOME II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Adjunct Professor, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA14979-06; R01DA014979 (NIH); DCNBR (Other: NIDA)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2015-07

CONDITIONS: Drug Use Disorders During Pregnancy
Keywords: pregnancy, opioid, cocaine, alcohol, benzodiazepines, neonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Usual RBT (t-RBT) (Active Comparator): Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach Social club Job club
  Interventions: Behavioral: Usual RBT (t-RBT)
- Reduced RBT (r-RBT) (Experimental): Individual therapy Skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach Social Club Job Club
  Interventions: Behavioral: Reduced RBT (r-RBT)
- Abbreviated RBT (a-RBT) (Experimental): Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Recreation
  Interventions: Behavioral: Abbreviated RBT (a-RBT); Behavioral: Early compliant r-RBT
- Enhanced RBT (e-RBT) (Active Comparator): Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach Social club Job club Recovery housing CAP short term housing admission Recovery sponsor
  Interventions: Behavioral: Enhanced RBT (e-RBT); Behavioral: Early non-compliant t-RBT
- Early compliant t-RBT (Active Comparator): r-RBT Individual therapy Skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach t-RBT: Social club Job club
  Interventions: Behavioral: Early compliant t-RBT
- Early non-compliant t-RBT (Active Comparator): t-RBT Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach Social club Job club e-RBT: Recovery housing CAP short term housing admission Recovery sponsor
  Interventions: Behavioral: Early non-compliant t-RBT; Behavioral: Early compliant r-RBT
- Early compliant r-RBT (Experimental): a-RBT Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Recreation r-RBT: Individual therapy Skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach
  Interventions: Behavioral: Abbreviated RBT (a-RBT); Behavioral: Early compliant r-RBT
- Early non-compliant r-RBT (Experimental): r-RBT Individual therapy Skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach t-RBT: Social Club Job Club
  Interventions: Behavioral: Early non-compliant t-RBT; Behavioral: Early non-compliant r-RBT

INTERVENTIONS:
Behavioral: Usual RBT (t-RBT) — Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach Social Club Job Club
  Arms: Usual RBT (t-RBT)
Behavioral: Reduced RBT (r-RBT) — Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach
  Arms: Reduced RBT (r-RBT)
Behavioral: Abbreviated RBT (a-RBT) — Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Recreation
  Arms: Abbreviated RBT (a-RBT); Early compliant r-RBT
Behavioral: Enhanced RBT (e-RBT) — Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach Social club Job Club Recovery housing CAP housing admission Recovery sponsor
  Arms: Enhanced RBT (e-RBT)
Behavioral: Early compliant t-RBT — r-RBT Individual therapy Skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach t-RBT: Social club Job club
  Arms: Early compliant t-RBT
Behavioral: Early non-compliant t-RBT — t-RBT Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach Social club Job club e-RBT: Recovery housing CAP short term housing admission Recovery sponsor
  Arms: Early non-compliant r-RBT; Early non-compliant t-RBT; Enhanced RBT (e-RBT)
Behavioral: Early compliant r-RBT — a-RBT Individual therapy CBT skills modules Functional assessment Behavior contracts Behavior graphing Recreation r-RBT: Individual therapy Skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach
  Arms: Abbreviated RBT (a-RBT); Early compliant r-RBT; Early non-compliant t-RBT
Behavioral: Early non-compliant r-RBT — r-RBT Individual therapy Skills modules Functional assessment Behavior contracts Behavior graphing Tangible rewards MI feedback Recreation Outreach t-RBT: Social Club Job Club
  Arms: Early non-compliant r-RBT

SUMMARY:
Objectives: This project is a Stage II behavioral development study designed to answer remaining critical questions necessary before disseminating Reinforcement Based Treatment (RBT) to the larger treatment community. These questions focus on the levels of intensity of RBT most efficacious for substance-using pregnant patients. Design: The proposed study utilizes a novel approach to conducting a controlled clinical trial, the sequential multiple assignment randomized trial (SMART) design. Participants (N=220) will first be randomized at treatment outset into either treatment-as-usual RBT or a reduced intensity RBT. All participants will receive a subsequent randomization based upon an assessment of their initial two weeks of treatment compliance. Early-non-compliant participants will be randomized to receive either the same or an increased level of RBT treatment intensity while early-compliant participants will be randomized to receive either the same or decreased level of treatment intensity and scope. Primary outcome measures include treatment completion, and maternal heroin, cocaine, and other illicit substance use. Secondary outcome measures include maternal measures of HIV risk behavior, and psychosocial functioning and neonatal measures of length of hospitalization, and birth outcomes. Significance: The proposed project's innovation includes: the novelty RBT, use of a cutting-edge SMART model, application of advanced statistical techniques and inclusion of a cost-effectiveness approach. The proposed project's significance is exceedingly high, as it will lay the foundation for later Stage III studies focused on dissemination of stepped care treatment programs for drug-addicted pregnant women that can be implemented not only in comprehensive care clinics but in diverse community settings that provide services to such women.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment entry at or before 34 weeks EGA with singleton fetus.
2. Evidence of opioid, cocaine and/or other primary illicit substance use.

Exclusion Criteria:

1. Severe medical or psychiatric concomitant condition interfering with treatment or needing hospitalization.
2. Age 17 years or younger.
3. Geographical constraints. These women are admitted only for a residential detoxification and often have plans to obtain aftercare in an outpatient or residential facility in closer proximity to their home. Thus, this greater distance from CAP increases the likelihood that these women will not return to CAP and will not deliver in a hospital that functions under similar protocols that operate in Baltimore City for treating drug-exposed neonates.

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Treatment Completion | Delivery (data extracted from medical record)
  Delivering a baby, regardless of delivery hospital, while enrolled in treatment.
Substance use | Once monthly until delivery and at six weeks post-partum
  Drug Use: Urinalysis testing and self reported use (days in past month) for opioids, cocaine and other illicit substance use.

SECONDARY OUTCOMES:
Alcohol | Once monthly until delivery and at six weeks post-partum
  Alcohol use: Urinalysis testing and self-reported (days in past month) of alcohol use
Maternal Obstetrical Course/Outcome | Delivery (data extracted from medical record)
  Available maternal data will be abstracted from the completed delivery record (i.e.., maternal urine toxicology results at delivery, complications during labor/delivery, placental abruption, type of delivery, maternal length of hospital stay).
Birth outcomes | Delivery (data extracted from medical record)
  Available birth outcome data will be extracted from infant medical records (i.e., birth weight, gestational age, infant complications).
Length of Hospital Stay | Upon release of infant from hospital (data extracted from medical record)
  Length of hospital stay is an indicator of health and well-being. The total days in the Newborn Nursery, Pediatrics and Neonatal Intensive Care will be abstracted from the medical records.
APGAR scores | Delivery (data extracted from medical record)
  Scores assigned at 1 and 5 minutes and any additional Apgar scoring if applicable will be extracted from the infant medical record

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Chisolm, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States